CLINICAL TRIAL: NCT06825247
Title: Assessment of the Psychosocial Sexual Health Competencies of Young Adults Born in France (including Those Whose Parents Were Born Abroad), and Proposal of a Sexual Health Promotion Model Adapted to the Needs Identified.
Acronym: ECOSSE
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Other Study IDs: CHM-2022/S10/16
Record Dates: First submitted 2025-02-10; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Sexual Health
Keywords: sexual health; psychosocial skills

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Young adults born in France and living in Pays de Loire

SUMMARY:
Every year, between 4,000 and 6,000 people discover their seropositivity to the human immunodeficiency virus (HIV). The dynamics of new discoveries vary according to sexual orientation and birthplace. MSM born in France show the sharpest improvement, while heterosexuals born in France show a more moderate decline, and intravenous drug users (IDUs) are still at a low ebb.

There is little fine-grained data available on a national scale to explain these dynamics among people living with HIV (PLHIV).

The acquisition of Psychosocial Competencies in sexual health is a prerequisite for good sexual health. It is important for all young people, and all the more so for young people from immigrant backgrounds, whom we hypothesize, despite the limited existing literature, to be more vulnerable due to the influence of their origins, their parents' culture or language barrier, or even religion.

The primary research question: What psychosocial skills should be included in a sexual health education program for young people born in France (including those born to migrant parents), to enable them to enjoy good sexual health in adulthood?

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 29 years
* Born in France or its territories,
* Be able to read and write French.

Exclusion Criteria:

* They are under guardianship,
* They refuse to take part in the study.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young adults born in France and living in Pays de Loire
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Health education models | from enrollment of first patient to end of all interviews (3 years)
  Design health education models adapted to the sexual health needs of young adults born in France and living in the Pays de Loire region

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Le Mans, Le Mans, France